CLINICAL TRIAL: NCT00788359
Title: Multi-center Trial to Validate Protein Biomarkers of a Pulmonary Exacerbation in Cystic Fibrosis
Brief Title: Cystic Fibrosis Foundation (CFF) Biomarkers of Exacerbation
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0366
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; pulmonary exacerbation; biomarkers
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (plasma)
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical and translational research in cystic fibrosis (CF) is hampered by a lack of biomarkers that can be used to identify promising new therapies. There is an urgent need for development and validation of biomarkers that more quickly predict the usefulness of potential drugs in CF and might prognosticate clinical course. In particular, combinations of protein biomarkers that can be obtained non-invasively offer great promise. The goal of this project is to determine whether protein biomarkers in blood can demonstrate a beneficial effect of treatment over two weeks. We intend to initially target an acute pulmonary exacerbation in CF because we know that subjects being treated with intravenous antibiotics and enhanced mucus clearance display clinical improvements within two weeks. We propose to prospectively collect blood samples from a large cohort of well-characterized CF persons serially during inpatient admissions for a pulmonary exacerbation and longitudinally during annual visits. Through this proposal, we hope to identify a CF lung injury biomarker panel that increases in the setting of an acute pulmonary exacerbation and improves rapidly following intravenous antibiotic therapy. Additionally, we will begin to explore whether this CF lung injury biomarker panel might also prognosticate clinical course including decline in pulmonary function. Finally, this study will serve as an important source of blood samples that will be banked for future biomarker and therapeutic studies designed to benefit the entire CF community.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as evidenced by a sweat chloride test >60mEq/L or by the presence of two known CF genetic mutations
* Male or female greater than or equal to 10 years of age
* Initiation of intravenous antibiotic therapy for a clinically diagnosed acute pulmonary exacerbation
* Ability to perform reproducible pulmonary function tests
* Willing to comply with the study procedures and willingness to provide written consent

Exclusion Criteria:

* Presence of a condition or abnormality that, in the opinion of the Principal Investigator (PI), would compromise the safety of the patient or quality of the data

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with CF greater than or equal to 10 years of age who are being started on intravenous (IV) antibiotics for a clinically diagnosed pulmonary exacerbation. Patients must demonstrate at least 3 of the 11 criteria for pulmonary exacerbation as defined by a Cystic Fibrosis Foundation (CFF) Consensus Conference. Treatment with a minimum of two IV antibiotics is required. We expect to enroll an approximately equal number of males and females. Most CF patients in our clinics are of white, non-Hispanic origin and we anticipate this ethnic mix to persist in this study. The majority of pediatric CF subjects will be admitted to the hospital for treatment purposes whereas many adults receive their IV antibiotics at home.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2007-12; Primary Completion 2012-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in concentration of individual protein biomarkers and various combinations of biomarkers in blood samples obtained pre and post IV antibiotic therapy | up to 21 days

SECONDARY OUTCOMES:
Changes in pulmonary function (particularly FEV1) measured by spirometry pre and post IV antibiotic therapy | Up to 21 days
Changes in bacterial densities (P. aeruginosa and other CF pathogens) in sputum samples obtained pre and post IV antibiotic therapy | Up to 21 days
Changes in serum white blood cell and absolute neutrophil counts obtained pre and post IV antibiotic therapy | Up to 21 days

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - National Jewish Medical and Research Center, Denver, Colorado
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Case Western Reserve University, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Heltshe SL, Goss CH, Thompson V, Sagel SD, Sanders DB, Marshall BC, Flume PA. Short-term and long-term response to pulmonary exacerbation treatment in cystic fibrosis. Thorax. 2016 Mar;71(3):223-9. doi: 10.1136/thoraxjnl-2014-206750. Epub 2015 Apr 24. PMID 25911223